CLINICAL TRIAL: NCT04321330
Title: An Open-Label, Single Arm, Multicenter Study to Investigate the Efficacy and Safety of Atezolizumab (Tecentriq) in Previously-Treated Patients With Advanced Thymic Carcinoma
Brief Title: A Study to Investigate the Efficacy and Safety of Atezolizumab (Tecentriq) in Previously-Treated Patients With Advanced Thymic Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41253
Record Dates: First submitted 2020-03-24; First posted 2020-03-25 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma, Thymic
MeSH Terms: conditions — Thymoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Participants will receive atezolizumab at a fixed dose of 1200 milligrams (mg) by intravenous (IV) infusion on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered by IV on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.
  Other Names: MPDL3280A; RO5541267; Tecentriq

SUMMARY:
This is a phase II, open-label, single-arm, multicenter study of the efficacy and safety of atezolizumab treatment in participants with advanced thymic carcinoma who failed prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of thymic carcinoma by the central pathology laboratory
* Advanced disease not amenable to curative treatment
* At least 1 prior line of chemotherapy
* Progression of disease must be documented prior to study entry
* Measurable disease, as defined by Response Evaluation Criteria for Solid Tumors, Version 1.1 (RECIST v1.1)
* Availability of a representative tumor specimen that is suitable for biomarkers research via central testing
* ECOG performance status 0 or1
* Life expectancy > 3 months
* Adequate hematologic and end-organ function within 14 days prior to the first study treatment
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* For women of childbearing potential: agreement to remain abstinent or use contraception

Exclusion Criteria:

* Disease which is amenable to radical treatment with surgery or radiation or a combination of treatments.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease within 3 months prior to initiation of study treatment unstable arrhythmia, or unstable angina.
* Prior treatment with chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered from adverse events due to a previously administered agent.
* Additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-07-16 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline up to approximately 3.5 years
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) on two consecutive occasions 4 weeks apart, as determined by the Investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Baseline up to approximately 3.5 years
  PFS is defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.
Overall Survival (OS) | Baseline up to approximately 3.5 years
  OS is defined as the time from initiation of study treatment to death from any cause.
Duration of Objective Response (DOR) | Baseline up to approximately 3.5 years
  DOR is defined as the time from initial response to disease progression or death among patients who have experienced a CR or PR (unconfirmed) during the study. Duration of response will be calculated based on disease status evaluated by the investigator according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline up to approximately 3.5 years
  DCR is defined as the proportion of patients who have a best overall response of CR or PR or SD, as determined by the investigator according to RECIST v1.1
Distribution of TMB Expression | Baseline up to approximately 3.5 years
  Positive is defined as >=10 Muts/Mb. Negative is defined as <10 Muts/Mb.
Distribution of PD-L1 Expression | Baseline up to approximately 3.5 years
  Positive is defined as TC or IC >=1%. Negative is defined as TC or IC <1%.
Percentage of Participants With Adverse Events | Baseline up to approximately 3.5 years
Percentage of Participants With Immune-Related Adverse Events | Baseline up to approximately 3.5 years

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University; Department of Breast, Chengdu
  - The Second Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - The affiliated hospital of Qingdao university, Qingdao
  - Shanghai Chest Hospital, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Remon J, Girard N, Novello S, de Castro J, Bigay-Game L, Bernabe R, Greillier L, Mosquera J, Cousin S, Juan O, Sampayo M, Besse B. PECATI: A Multicentric, Open-Label, Single-Arm Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab and Lenvatinib in Pretreated B3-Thymoma and Thymic Carcinoma Patients. Clin Lung Cancer. 2022 May;23(3):e243-e246. doi: 10.1016/j.cllc.2021.07.008. Epub 2021 Jul 20. PMID 34393061